CLINICAL TRIAL: NCT02808455
Title: A Phase 1, Open-Label, Single-Dose, Randomized, 2-Period, 2-Treatment-Sequence Crossover Study to Assess the Relative Bioavailability of Pacritinib Following Oral Administration as Capsule and Solution Formulations in Healthy Subjects
Brief Title: Study to Assess the Relative Bioavailability of Pacritinib Following Oral Administration as Capsule and Solution Formulations in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CTI BioPharma (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PAC101
Record Dates: First submitted 2016-05-03; First posted 2016-06-21 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2016-06

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — 11-(2-pyrrolidin-1-ylethoxy)-14,19-dioxa-5,7,26-triazatetracyclo(19.3.1.1(2,6).1(8,12))heptacosa-1(25),2(26),3,5,8,10,12(27),16,21,23-decaene; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sequence I: A/B (Experimental): Treatment A: pacritinib 400 mg capsule
  Interventions: Drug: (Treatment A); Drug: (Treatment B)
- Sequence II: B/A (Experimental): Treatment B: pacritinib 80 mg solution
  Interventions: Drug: (Treatment A); Drug: (Treatment B)

INTERVENTIONS:
Drug: (Treatment A) — Four 100-mg capsules of pacritinib administered as a single oral dose
  Other Names: Pacritinib 400 mg Capsule
Drug: (Treatment B) — A single 80-mg oral solution dose of pacritinib
  Other Names: Pacritinib 80 mg Solution

SUMMARY:
This was a randomized, 2-period, 2-treatment-sequence crossover study to determine the relative bioavailability of pacritinib following administration as a 400 mg oral dose of four 100 mg pacritinib capsules and an 80 mg dose of an oral solution and to characterize the PK and major human metabolites of pacritinib.

DETAILED DESCRIPTION:
Twelve healthy subjects will be enrolled in the study (6 subjects per sequence) at a single clinical site with the intent that 12 subjects complete Periods 1 and 2 in the study. Subjects will be randomly assigned to 2 possible sequences (6 subjects per sequence) on Day 1 of Period 1. Subjects will be randomly assigned to 2 possible sequences. Each subject received 2 treatments (a 400 mg oral dose of four 100 mg pacritinib capsules and an 80 mg oral solution dose of pacritinib) in a 2-period crossover design. Each treatment will be administered as monotherapy during 1 of 2 treatment periods with a 7-day washout period between administrations of each study medication.

ELIGIBILITY:
Inclusion Criteria:

1. males or females, between 18 and 55 years of age, inclusive;
2. BMI between 18.5 and 32.0 kg/m2, inclusive;
3. in good health, determined by no clinically significant findings from medical history, physical examination, and vital signs;
4. normal 12-lead ECG or ECG findings (including RR, PR, and QT intervals; QT interval corrected using Fridericia's formula [QTcF]; QRS duration; and ventricular heart rate) deemed not clinically significant;
5. clinical laboratory evaluations (including clinical chemistry panel [fasted at least 10 hours], CBC, and UA) within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator in consultation with the Sponsor;
6. negative test for selected drugs of abuse (including alcohol) at Screening and at Check-in (Day -1 of Period 1);
7. negative hepatitis panel (including HBsAg and anti-HCV) and negative HIV antibody screens;
8. females of childbearing potential must be non-pregnant and non-lactating, and agree to use one of the following forms of contraception from the time of signing the informed consent or 10 days prior to Check-in (Day -1) of Period 1 until 30 days after the final dose administration: non-hormonal intrauterine device (IUD) with spermicide; female condom with spermicide; contraceptive sponge with spermicide; intravaginal system (eg, NuvaRing®); diaphragm with spermicide; cervical cap with spermicide; male sexual partner who agrees to use a male condom with spermicide; sterile sexual partner; or abstinence. Oral, implantable, transdermal, or injectable hormonal contraceptives may not be used from the time of signing the informed consent or 10 days prior to Check-in (Day -1) of Period 1 until 14 days after the final dose administration. For all females, the pregnancy test result must be negative at Screening and Check-in (Day -1) of Period 1. Females not of childbearing potential must be postmenopausal for at least 1 year or surgically sterile (eg, tubal ligation, hysterectomy) for at least 90 days;
9. males will be surgically sterile (ie, vasectomy, documented in the medical record by a physician) or agree to use, from Check-in (Day -1) of Period 1 until 90 days following Study Completion/ET, 1 of the following approved methods of contraception: male condom with spermicide; sterile sexual partner; or use by female sexual partner of an IUD with spermicide, a female condom with spermicide, a contraceptive sponge with spermicide, an intravaginal system, a diaphragm with spermicide, a cervical cap with spermicide, or oral, implantable, transdermal, or injectable contraceptives. Subjects must agree to refrain from sperm donation from Check-in (Day -1) of Period 1 until 90 days following Study Completion/ET;
10. able to comprehend and willing to sign an Informed Consent Form (ICF).

Exclusion Criteria:

1. prior ingestion of pacritinib;
2. history or clinical manifestation of clinically significant cardiovascular, pulmonary, hepatic (eg, hepatitis), renal, hematologic, gastrointestinal (eg, celiac disease, peptic ulcer, gastroesophageal reflux, inflammatory bowel disease), metabolic, allergic, dermatological, neurological, or psychiatric disorder (as determined by the Investigator in consultation with the Sponsor; appendectomy and cholecystectomy are not considered to be clinically significant events);
3. significant abnormalities in liver function tests (alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase >1.5 × upper limit of normal [ULN]; gamma-glutamyl transferase >2 × ULN; or total bilirubin >1.3 × ULN) or kidney function tests (serum creatinine > ULN) that are considered clinically significant by the Investigator, in consultation with the Sponsor;
4. history of malignancy, except the following: cancers determined to be cured or in remission for ≥5 years, curatively resected basal cell or squamous cell skin cancers, cervical cancer in situ, or resected colonic polyps;
5. history of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator in consultation with the Sponsor;
6. history of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs except that appendectomy, cholecystectomy, and hernia repair will be allowed;
7. history of Gilbert's Syndrome;
8. history or presence of ECG QTcF >450 msec, factors that increase risk for QTc interval prolongation (eg, heart failure, hypokalemia [defined as serum potassium <3.0 mEq/L that is persistent and refractory to correction], or family history of long QT interval syndrome);
9. history of alcoholism or drug addiction within 1 year prior to Check-in (Day -1) of Period 1;
10. use of tobacco- or nicotine-containing products within 6 months prior to Check-in (Day -1) of Period 1 and during the entire study;
11. consumption of alcohol- or caffeine-containing foods and beverages for 72 hours prior to Screening and during the entire study;
12. consumption of grapefruit-containing foods and beverages or other CYP3A4 inhibitors or inducers for 72 hours prior to Screening and during the entire study. A list of CYP3A4 inhibitors and inducers is provided in;
13. subjects will refrain from strenuous exercise from 48 hours prior to Check-in (Day -1) of Period 1 and during the period of confinement at the CRU and will otherwise maintain their normal level of physical activity throughout the entire study (ie, will not begin a new exercise program nor participate in any unusually strenuous physical exertion);
14. participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives or 30 days prior to Check-in (Day -1) of Period 1, whichever is longer, and during the entire study;
15. female subjects who are unable to refrain from the use of oral, implantable, injectable, or transdermal hormonal contraceptives within 10 days prior to Check-in (Day -1) of Period 1 or from the time of signing the informed consent until 14 days after the final dose administration;
16. use of any prescription medications and/or products within 14 days prior to Check-in (Day -1) of Period 1 and during the entire study, unless deemed acceptable by the Investigator in consultation with the Sponsor;
17. use of any over-the-counter, non-prescription medications (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within 7 days prior to Check-in (Day -1) of Period 1 and during the entire study, unless deemed acceptable by the Investigator in consultation with the Sponsor;
18. poor peripheral venous access;
19. donation of blood from 30 days prior to Screening through Study Completion/ET, inclusive, or plasma from 2 weeks prior to Screening through Study Completion/ET, inclusive;
20. receipt of blood products within 2 months prior to Check-in (Day -1) of Period 1;
21. any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  For each subject, the following PK parameters were calculated, whenever possible, based on the plasma concentrations of pacritinib and pacritinib M1 metabolite, using noncompartmental methods.
The area under the plasma concentration-time curve from time zero to time of the last measured concentration above the limit of quantification (AUC0-t) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  For each subject, the following PK parameters were calculated, whenever possible, based on the plasma concentrations of pacritinib and pacritinib M1 metabolite, using noncompartmental methods.
The time to reach maximum plasma concentration (tmax) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  For each subject, the following PK parameters were calculated, whenever possible, based on the plasma concentrations of pacritinib and pacritinib M1 metabolite, using noncompartmental methods.
The area under the plasma concentration-time curve from zero to infinity (AUC0-∞) | Plasma: 0, 1, 2, 4, 6, 8, 12, 24, 36, 48, 60, 72, 84, 96, 108, 120, 144, and 168 hrs post-dose
  For each subject, the following PK parameters were calculated, whenever possible, based on the plasma concentrations of pacritinib and pacritinib M1 metabolite, using noncompartmental methods.
Area under the effect-time curve from Hour 0 to the last measurable activity level | Blood samples were collected up to 168 hours post pacritinib dose
  For each subject, the following PD parameters were calculated, whenever possible, based on the stimulated pSTAT3/unstimulated Total STAT3 ratio in PBMCs, using noncompartmental methods

SECONDARY OUTCOMES:
Treatment emergent adverse events | Day 1 to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Hugh Coleman, DO, Principal Investigator — Covance Clinical Research Unit
Locations (1):
- Covance Clinical Research Unit, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes